CLINICAL TRIAL: NCT06317220
Title: Vedolizumab for the Treatment of Collagenous Gastritis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Takeda (Industry)
Responsible Party: Principal Investigator, Michael Dougan, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000152
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Collagenous Gastritis
Keywords: collagenous gastritis, vedolizumab
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vedolizumab 300mg (Experimental): * Dose: 300mg
  * Administration: Intravenous (IV)
  * Frequency: Weeks 0, 2, 6, and then every 8 weeks
  * Duration: 54 weeks (1 year)
  Interventions: Biological: Vedolizumab

INTERVENTIONS:
Biological: Vedolizumab — Administered over 30 minute infusion at MGH main campus
  Other Names: Entyvio

SUMMARY:
The goal of this clinical trial is to learn about how vedolizumab may affect patients with collagenous gastritis (CG). The main questions it aims to answer are:

* Whether vedolizumab can reduce CG symptoms
* Whether vedolizumab is safe to take for patients with CG

Participants in this study will:

* Receive vedolizumab through an IV ("infusion")
* Complete a survey at each infusion visit
* Have blood collected at each infusion visit
* Undergo an endoscopy with biopsy at 2 timepoints

DETAILED DESCRIPTION:
Eligible participants will receive vedolizumab through an IV ("infusion") at week 0, then week 2, then week 6. Participants who respond well to the treatment after the first 3 infusions and are interested in continuing will receive vedolizumab every 8 weeks for about 1 year. At each visit, participants will be asked about their collagenous gastritis symptoms and any changes in their health or medications.

Blood samples will be collected from participants at every vedolizumab infusion. Some of these samples will be collected for safety purposes, some will be collected to monitor CG progression, and some will be collected for research purposes.

During the screening period and a few months after beginning treatment, the study doctor will perform an upper endoscopy to help determine whether vedolizumab has improved each participant's CG. An upper endoscopy is a procedure where the doctor inserts a small tube with a camera through the mouth and down the throat to look at the upper gastrointestinal tract (the esophagus, stomach, and part of the small intestine). During the procedure, biopsies will be collected to monitor CG and for research purposes. All participants will be given medication to make them comfortable throughout the duration of the procedure, which lasts approximately 10 to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 or older
* Weight of at least 40kg
* Has a biopsy-confirmed diagnosis of collagenous gastritis
* Agrees to all required study procedures
* Presence of one or more collagenous gastritis symptom at a severity of Grade 1 or higher at the time of enrollment: abdominal pain, nausea, diarrhea, bloating, vomiting, flatulence, constipation, fatigue, headache, rash

Exclusion Criteria:

* Unable to independently provide informed consent or assent
* Allergic to vedolizumab or any of its components

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in symtpoms | 12 Weeks
  Change in symptoms associated with collagenous gastritis after 12 weeks of vedolizumab treatment, measured via patient-reported symptom questionnaire scores collected at each visit. Response is defined as a decrease of at least 1 Grade (DAIDS) in the most severe symptom reported at baseline. Surveys will be scored from 0 to 38, with higher scores indicating more severe symptoms and lower outcomes indicating no symptoms or more mild symptoms.

SECONDARY OUTCOMES:
Response durability | 54 Weeks
  Durability of symptomatic response to vedolizumab over the first year of treatment will be measured via patient-reported symptom questionnaire scores collected at each visit. Surveys will be scored from 0 to 38, with higher scores indicating more severe symptoms and lower outcomes indicating no symptoms or more mild symptoms.
Histologic response | 12 weeks (+/- 4 weeks)
  Histologic response to vedolizumab will be assessed by comparing gastric histology from on-treatment biopsies and, if available, compared to baseline (within 1 year) gastric histology
Incidence of treatment-emergent adverse events (safety) | 54 Weeks
  Safety will be assessed by adverse event (AE) rates throughout the first year of treatment. Severity will be graded according to the DAIDS grading table (v2.1).

OTHER OUTCOMES:
Immunologic response in gastric mucosa | 54 Weeks
  Immunologic response in the gastric mucosa will be assessed via flow cytometry and scRNA-seq of gastric biopsies and, if available, compared to baseline (within 1 year) gastric biopsies
Immunologic response in peripheral blood | 54 Weeks
  Immunologic response in peripheral blood will be assessed via flow cytometry and scRNA-seq of peripheral blood mononuclear cells as well as serum proteomics

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States